CLINICAL TRIAL: NCT06421181
Title: Hemodynamic Effects of Anesthesia Induction
Acronym: KEM-HEN
Status: Recruiting | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: KEM-HEN
Record Dates: First submitted 2024-04-26; First posted 2024-05-20 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Patients Undergoing Anaesthesia Induction
Keywords: Hemodynamic monitoring; Point-of-care ultrasound; Point-of-care echocardiography; Anaesthesia induction; Respiratory effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The idea of that project is to characterize the hemodynamic changes of a daily used clinical intervention (induction of anesthesia) in a highly controlled environment by two hemodynamic monitoring devices. The aim is an advanced hemodynamic profiling of this intervention and additionally screen for changes in flow patterns in an exploratory fashion.

Both devices complement one another in their hemodynamic profiling ability. One device is a continuous monitoring with instant traceable changes and the other an intermittent point-of-care ultrasound/echocardiography device with advanced possibilities for differential diagnostics.

A second purpose is to test the possibility to implement advanced echocardiography in a point-of-care approach during anaesthesia induction and evaluate the time and quality of a comprehensive analysis by a not-certified anaesthetists with an echocardiography device with features of artificial intelligence versus a certified expert.

DETAILED DESCRIPTION:
Mortality after surgery is still high and high-risk procedures are associated to high postoperative complication rates. For hemodynamic monitoring, a meta-analysis showed a reduction in mortality and especially for the esophageal Doppler a reduction in postoperative complications. However, the effects reducing mortality and morbidity have to be considered as low. Probably, this is the reason why daily clinical implementation rates of hemodynamic monitoring are low, too.

However, hemodynamic studies only focus on intraoperative optimization, but recent publications suggested that taking preoperative individual hemodynamic values for arterial blood pressure and cardiac index as targets for optimization provides advanced therapeutic options. Lastly, both studies do not provide data about the preoperative values and their changes during the induction of anesthesia.

Our own data confirm that the induction of anesthesia, the establishment of a working epidural and the surgical incision of the abdomen leads to decreased cardiac index and markers of inotropy in otherwise cardiovascular healthy patients. However, the intervention studies and our own data strongly suggest that starting hemodynamic monitoring after the induction of anesthesia or the surgical incision may foreclose that the clinician can guide the hemodynamic therapy towards individualized goals. Additionally, the corrective treatment in this scenario could be different from just vasopressors.

Nevertheless, in contrast to our own data a recent study showed that hypotension in the post-induction period is primarily associated with a decreased vascular tone due to anesthetic agents, suggesting that the appropriate treatment is vasopressors.

A detailed hemodynamic profiling of non-cardiac patients undergoing high-risk cancer surgery prior, during and after the induction of anaesthesia may provide new insights about the effects of anaesthetic drugs, positive pressure ventilation, and changes of sympathetic tone.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparotomy in the hospital Evangelische Kliniken Essen-Mitte
* Due to the invasiveness of the planned surgery there is an indication for an arterial and central-venous line as well as an peridural catheter

Exclusion Criteria:

* Age < 18 years
* Lack of written informed consent
* Insufficient language skills
* Unwillingness to have pseudonymized disease data stored at the study site and lack of consent to share anonymized data as part of the clinical trial
* American society of anaesthesiologists physical status higher as grade 3
* congestive heart failure with a grade of 2 or higher according to the New York heart association (NYHA)
* Ischemic cardiopathy with a grade of 2 or higher according to the Canadian cardiovascular society (CCS)
* Known severe valve pathologies of the heart
* Chronic kidney disease with dependency of hemodialysis
* Atrial fibrillation ora trail flutter
* Pulmonary hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of advanced primary ovarian cancer will be screened prior to cytoreductive surgery in cooperation with the colleagues of gynaecological oncology. If the patients are eligible they will be informed to give consent.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change of heart rate assessed in percentages during the induction of anaesthesia | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The heart rate will be monitored continuously to detect any change of it during the induction of anaesthesia. The change will be described in percentages.
Longitudinal change of arterial blood pressure assessed in percentaqes during the induction of anaesthesia | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The arterial blood pressures will be monitored continuously to detect any change of it during the induction of anaesthesia. The change will be described in percentages.
Longitudinal change of stroke volume assessed in percentaqes during the induction of anaesthesia | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The stroke volume will be monitored continuously to detect any change of it during the induction of anaesthesia. The change will be described in percentages.
Longitudinal change of myocardial strain imaging assessed by transthoracic echocardiography during the induction of anaesthesia | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The echocardiographic feature of strain imaging for the analysis of contractile performance of the myocardium will be monitored prior to induction and after induction of anaesthesia to detect any changes

SECONDARY OUTCOMES:
Changes in percentages in a comprehensive echocardiographic assessment of the right ventricle and atrium | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The echocardiographic features will be monitored prior to induction and after induction of anaesthesia to detect any changes
Changes of the left ventricular and atrial volume in percentages assessed by a transthoracic echocardiography | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The echocardiographic parameter will be monitored prior to induction and after induction of anaesthesia to detect any changes.
Changes of the left ventricular systolic and diastolic function in percentages assessed by a transthoracic echocardiography | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The echocardiographic features will be monitored prior to induction and after induction of anaesthesia to detect any changes
Changes of function of the cardiac valves assessed by a transthoracic echocardiography | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The echocardiographic features will be monitored prior to induction and after induction of anaesthesia to detect any changes of the cardiac valve functions like increase of regurgitation
Changes in percentage of the cardiocirculatory flow in an advanced hemodynamic monitoring device based on a pulse-contour methodology in a continuous fashion during induction of anaesthesia | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The haemodynamic features will be monitored prior to the start of induction up to the end of induction of anaesthesia to detect any changes
Changes of flow profiles of the splanchnic vessels as well as peripheral arteries determined by ultrasound | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The ultrasound features will be monitored prior to induction and after induction of anaesthesia to detect any changes
Mean systemic filling pressure (MSFP) | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  The MSFP will be determined based on the stop-flow-methodology to determine additionally venous return characteristics
Baroreceptor sensitivity (BRS) | Time from the start of anaesthesiological monitoring up to start of surgical measures, up to four hours
  BRS will be determined to analyse the impact of drugs of anaesthesia induction on the vegetative nervous system. The assessment is based on invasive measurement of the arterial blood pressure in combination with the electrocardiogram

OTHER OUTCOMES:
Examination times of the echocardiographic assessment by a not-certified expert | Time from the start of anaesthesiological monitoring up to the start of anaesthesia induction, up to four hours
  The characteristics of an echocardiographic assessment will be analysed to examine the feasibility within clinical routine and the results will be compared to the results of a certified echocardiographic expert
Implementation rates in percentages of the echocardiographic assessment by a not-certified expert during clinical care | Time from the start of anaesthesiological monitoring up to the start of anaesthesia induction, up to four hours
  The characteristics of an echocardiographic assessment will be analysed to examine the feasibility within clinical routine and the results will be compared to the results of a certified echocardiographic expert
Number of missed diagnositics of the echocardiographic assessment by a not-certified expert vs. an assessment by a certified examiner | Time from the start of anaesthesiological monitoring up to the start of anaesthesia induction, up to four hours
  The characteristics of an echocardiographic assessment will be analysed to examine the feasibility within clinical routine and the results will be compared to the results of a certified echocardiographic expert
Incidence and description of postoperative complications | Time of hospital stay, i.d. from the time of surgery up to discharge from the hospital, up to 30 days after surgery
  The complications will be graded according to the "Clavien-Dindo" classification from one to five with one being a minor complication and five being death
Incidence and description of postoperative organ dysfunctions | Time of hospital stay, i.d. from the time of surgery up to discharge from the hospital, up to 30 days after surgery
  The incidence of organ dysfunctions will be based on laboratory results and or pathophysiological features like delayed bowel opening after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aarne Feldheiser, M.D., PhD., Principal Investigator — Evangelische Kliniken Essen-Mitte
Locations (1):
- Evangelische Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chong MA, Wang Y, Berbenetz NM, McConachie I. Does goal-directed haemodynamic and fluid therapy improve peri-operative outcomes?: A systematic review and meta-analysis. Eur J Anaesthesiol. 2018 Jul;35(7):469-483. doi: 10.1097/EJA.0000000000000778. PMID 29369117
- [Background] Ripolles-Melchor J, Casans-Frances R, Espinosa A, Abad-Gurumeta A, Feldheiser A, Lopez-Timoneda F, Calvo-Vecino JM; EAR Group, Evidence Anesthesia Review Group. Goal directed hemodynamic therapy based in esophageal Doppler flow parameters: A systematic review, meta-analysis and trial sequential analysis. Rev Esp Anestesiol Reanim. 2016 Aug-Sep;63(7):384-405. doi: 10.1016/j.redar.2015.07.009. Epub 2016 Feb 10. English, Spanish. PMID 26873025
- [Background] Sessler DI, Bloomstone JA, Aronson S, Berry C, Gan TJ, Kellum JA, Plumb J, Mythen MG, Grocott MPW, Edwards MR, Miller TE; Perioperative Quality Initiative-3 workgroup; POQI chairs; Miller TE, Mythen MG, Grocott MP, Edwards MR; Physiology group; Preoperative blood pressure group; Intraoperative blood pressure group; Postoperative blood pressure group. Perioperative Quality Initiative consensus statement on intraoperative blood pressure, risk and outcomes for elective surgery. Br J Anaesth. 2019 May;122(5):563-574. doi: 10.1016/j.bja.2019.01.013. Epub 2019 Feb 27. PMID 30916004
- [Background] Kouz K, Wegge M, Flick M, Bergholz A, Moll-Khosrawi P, Nitzschke R, Trepte CJC, Krause L, Sessler DI, Zollner C, Saugel B. Continuous intra-arterial versus intermittent oscillometric arterial pressure monitoring and hypotension during induction of anaesthesia: the AWAKE randomised trial. Br J Anaesth. 2022 Oct;129(4):478-486. doi: 10.1016/j.bja.2022.06.027. Epub 2022 Aug 23. PMID 36008202
- [Background] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220
- [Background] Nicklas JY, Diener O, Leistenschneider M, Sellhorn C, Schon G, Winkler M, Daum G, Schwedhelm E, Schroder J, Fisch M, Schmalfeldt B, Izbicki JR, Bauer M, Coldewey SM, Reuter DA, Saugel B. Personalised haemodynamic management targeting baseline cardiac index in high-risk patients undergoing major abdominal surgery: a randomised single-centre clinical trial. Br J Anaesth. 2020 Aug;125(2):122-132. doi: 10.1016/j.bja.2020.04.094. PMID 32711724
- [Background] Saugel B, Bebert EJ, Briesenick L, Hoppe P, Greiwe G, Yang D, Ma C, Mascha EJ, Sessler DI, Rogge DE. Mechanisms contributing to hypotension after anesthetic induction with sufentanil, propofol, and rocuronium: a prospective observational study. J Clin Monit Comput. 2022 Apr;36(2):341-347. doi: 10.1007/s10877-021-00653-9. Epub 2021 Feb 1. PMID 33523352
- [Result] Middel C, Stetzuhn M, Sander N, Kalkbrenner B, Tigges T, Pielmus AG, Spies C, Pietzner K, Klum M, von Haefen C, Hunsicker O, Sehouli J, Konietschke F, Feldheiser A. Perioperative advanced haemodynamic monitoring of patients undergoing multivisceral debulking surgery: an observational pilot study. Intensive Care Med Exp. 2023 Sep 8;11(1):61. doi: 10.1186/s40635-023-00543-1. PMID 37682496
- [Result] Feldheiser A, Juhl-Olsen P, Nordine M, Stetzuhn M, Wiegank L, Knebel F, Treskatsch S, Berger C. A comprehensive echocardiographic analysis during simulated hypovolaemia: An observational study. Eur J Anaesthesiol. 2023 Aug 1;40(8):578-586. doi: 10.1097/EJA.0000000000001863. Epub 2023 Jun 1. PMID 37265333